CLINICAL TRIAL: NCT00826462
Title: Physiotherapy Alone, in Combination With Corticosteroid Injection or Wait-and-see for Acute Lateral Epicondylitis in General Practice: a Randomised, Placebo-controlled Study With 12 Months Follow-up
Brief Title: Treatment Study of Steroid Injection and Physical Therapy for Acute Lateral Epicondylitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Allmennmedisinsk forskningsfond, Norway (Unknown)
Responsible Party: Principal Investigator, Morten Lindbaek, Professor Dr.med, University of Oslo
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006-002283-26
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Results first posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-11

CONDITIONS: Tennis Elbow; Epicondylitis, Lateral Humeral
Keywords: Randomised; Placebo-controlled; double blind; Intervention study; Primary health care
MeSH Terms: conditions — Tennis Elbow | interventions — Triamcinolone; Lidocaine; Sodium Chloride; Physical Therapy Modalities; Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Corticosteroid injection in combination with physical therapy
  Injection with triamcinolone 10 mg and 10 mg of lidocaine at start and at 3 weeks in combination with physiotherapy for 6 weeks (12 treatments with deep friction massage, Mill's manipulation, soft tissue treatment and home exercises) Naprosyn Entero 500 mg bid for 14 days
  Interventions: Drug: triamcinolone; Drug: Lidocaine; Other: Physiotherapy; Drug: Naproxen
- 2 (Placebo Comparator): Placebo injection in combination with physical therapy
  Injection with sodium chloride and 10 mg of lidocaine at start and at 3 weeks in combination with physiotherapy for 6 weeks (12 treatments with deep friction massage, Mill's manipulation, soft tissue treatment and home exercises) Naprosyn entero 500 mg bid for 14 days
  Interventions: Drug: Placebo; Drug: Lidocaine; Other: Physiotherapy; Drug: Naproxen
- 3 (Active Comparator): Control group: wait-and-see treatment Naprosyn entero 500 mg bid for 14 days
  Interventions: Drug: Naproxen

INTERVENTIONS:
Drug: triamcinolone — Injection with triamcinolone 10 mg at start and at 3 weeks
  Other Names: Kenacort - T (triamcinolone); Xylocaine (lidocaine)
  Arms: 1
Drug: Placebo — Injection with sodium chloride at start and at 3 weeks
  Other Names: Sodium chloride
  Arms: 2
Drug: Lidocaine — 10 mg of lidocaine at start and at 3 weeks
  Other Names: Xylocaine
  Arms: 1; 2
Other: Physiotherapy — 12 treatments with deep friction massage, Mill's manipulation, soft tissue treatment and home exercises
  Other Names: Physical therapy
  Arms: 1; 2
Drug: Naproxen — Naproxen 500 mg bid for 14 days
  Other Names: Naprosyn entero

SUMMARY:
The purpose of this study is to compare the clinical effect of physiotherapy alone or combined with corticosteroid injection in the initial treatment of lateral epicondylitis in a primary care setting.

To find the short and long term effect of physiotherapy with Mill's manipulation, deep friction massage and exercise therapy.

To ascertain wether the outcome is influenced by corticosteroid injection, which has been shown to be of benefit alone in the short term?

DETAILED DESCRIPTION:
Much has been written about lateral epicondylitis/tennis elbow reflecting the existence of many treatments for the condition. However, there is no consensus as to which treatment gives the best results.

Based on the latest meta-studies and reviews from the Cochrane Library, one may conclude that there is evidence of a short-term effect of topical or per oral NSAIDs. The same is true for manipulation and exercise. Corticosteroid injection has also been shown to have short-term effect, but not beyond 6 weeks. Ultrasound has a possible short-term effect based on one meta-analysis. Extra corporeal shock wave therapy does not seem to be effective. The treatment with acupuncture, orthosis, surgery or long-term NSAIDs has no support in the literature, and it is impossible to draw any conclusions about the effects or absence thereof. In fact, there is scant support for any long-term treatment in the literature.

We have found two studies to be of special interest (see citations below). Both have been done in a primary care setting with one-year follow up. One study compares corticosteroid injection with physical therapy (ultrasound, manipulation and exercise) and a wait-and-see group. The other compares corticosteroid injection with naproxen orally and placebo-medication. Both conclude that corticosteroid injection is a safe and effective treatment as pain-relief during the first 6 weeks, and that the effect of this treatment is better than physical therapy, wait-and-see and naproxen orally within the same time-frame. Physical therapy in one study gives some, but not statistically significantly better long-term (one year) effect than wait-and-see treatment.

There seems to be some indication that corticosteroid injection is a good alternative for the first 6 weeks. We find there is a good reason to investigate the long-term effects of physical therapy. At the same time, it would be interesting to see whether the good initial response from corticosteroid injection may be extended if combined with physiotherapy.

This randomised, placebo-controlled study will be conducted in general practice in the town of Sarpsborg, Ostfold County, Norway including patient aged 18-70 years with pain of recent onset from the lateral part of the elbow. After a treatment-period of 6 weeks, the patient is followed for a total of 12 months.

Patients are recruited by interested general practitioners in the city of Sarpsborg and surroundings and remitted to two study-physicians who make the initial evaluation of inclusion- and exclusion criteria, as well as treatment, follow-up and outcome assessments during the whole study-period. The patients are treated by one of the two study-physicians in the 6-weeks treatment-period. From the 6. week, the patient sees the other physician, who is unaware of the allocated intervention, for further registration and assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Pain from the lateral part of the elbow
* The pain increases on resisted dorsiflexion of the wrist with the elbow extended and the fingers flexed or the pain increases on resisted radial deviation of the wrist or the pain increases on resisted extension of the 3. finger

Exclusion Criteria:

* Duration of complaints less than 2 weeks or more than 3 months
* The tenderness is located within the muscle body itself in the proximal part of the short radial extensors muscle of the wrist (Cyriax type IV)9.
* Treatment within the last 12 months for the same condition with corticosteroid injection or physiotherapy
* Bilateral complaints
* Previous surgical treatment for lateral epicondylitis
* Deformities of the elbow (congenital or acquired)
* Cervical radiculopathy or referred pain from neck or shoulder
* Previous fractures or tendon ruptures in the elbow
* Systemic musculoskeletal disease
* Previous allergic reactions to corticosteroids or lidocaine
* Contraindications to corticosteroids or NSAIDs:

  * On-going or previous gastro-intestinal bleeding
  * previous ulcer or dyspepsia, severe asthma
  * on-going systemic infection
  * local skin-infection
  * recently vaccinated with live virus
  * coagulopathies
  * systemic lupus erythematodes
  * severe liver- or kidney-disease
  * heart failure
  * diabetes
  * use of warfarin or NSAIDS
* Pregnancy or breast-feeding
* Fertile females not on effective birth control
* Psycho-social or other reasons for not being able to participate throughout the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2009-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morten Lindbaek, Ph. D., Study Chair — University of Oslo
Locations (1):
- Grålum legesenter, Sarpsborg, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Olaussen M, Holmedal O, Mdala I, Brage S, Lindbaek M. Corticosteroid or placebo injection combined with deep transverse friction massage, Mills manipulation, stretching and eccentric exercise for acute lateral epicondylitis: a randomised, controlled trial. BMC Musculoskelet Disord. 2015 May 20;16:122. doi: 10.1186/s12891-015-0582-6. PMID 25989985
- [Derived] Holmedal O, Olaussen M, Mdala I, Natvig B, Lindbaek M. Predictors for outcome in acute lateral epicondylitis. BMC Musculoskelet Disord. 2019 Aug 17;20(1):375. doi: 10.1186/s12891-019-2758-y. PMID 31421668
- [Derived] Olaussen M, Holmedal O, Lindbaek M, Brage S. Physiotherapy alone or in combination with corticosteroid injection for acute lateral epicondylitis in general practice: a protocol for a randomised, placebo-controlled study. BMC Musculoskelet Disord. 2009 Dec 4;10:152. doi: 10.1186/1471-2474-10-152. PMID 19961603

RESULTS

PARTICIPANT FLOW:
Groups:
- Corticosteroid Injection in Combination With Physical Therapy: Corticosteroid injection in combination with physical therapy
  Injection with triamcinolone 10 mg and 10 mg of lidocaine at start and at 3 weeks in combination with physiotherapy for 6 weeks (12 treatments with deep friction massage, Mill's manipulation, soft tissue treatment and home exercises) Naprosyn Entero 500 mg bid for 14 days
  triamcinolone: Injection with triamcinolone 10 mg at start and at 3 weeks
  Lidocaine: 10 mg of lidocaine at start and at 3 weeks
  Physiotherapy: 12 treatments with deep friction massage, Mill's manipulation, soft tissue treatment and home exercises
  Naproxen: Naproxen 500 mg bid for 14 days
- Placebo Injection in Combination With Physical Therapy: Placebo injection in combination with physical therapy
  Injection with sodium chloride and 10 mg of lidocaine at start and at 3 weeks in combination with physiotherapy for 6 weeks (12 treatments with deep friction massage, Mill's manipulation, soft tissue treatment and home exercises) Naprosyn entero 500 mg bid for 14 days
  Placebo: Injection with sodium chloride at start and at 3 weeks
  Lidocaine: 10 mg of lidocaine at start and at 3 weeks
  Physiotherapy: 12 treatments with deep friction massage, Mill's manipulation, soft tissue treatment and home exercises
  Naproxen: Naproxen 500 mg bid for 14 days
- Control Group: Wait-and-see Treatment: Control group: wait-and-see treatment Naprosyn entero 500 mg bid for 14 days
  Naproxen: Naproxen 500 mg bid for 14 days
Period: Overall Study
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Started | 59 | 58 | 60
Completed | 52 | 53 | 52
Not Completed | 7 | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment | Total
Number analyzed (Participants) | 59 | 58 | 60 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (9.6) | 48.8 (9.4) | 44.0 (9.7) | 46.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 20 | 25 | 71
  Male | 33 | 38 | 35 | 106
Region of Enrollment [Number; unit: participants]
  Norway | 59 | 58 | 60 | 177

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success - Event Rates in Each Group
Description: Unadjusted event rates of treatment success, defined as participants rating themselves 'much improved' or 'completely recovered' on a six point scale. Percentage with 99% confidence interval.
Time Frame: 6 - 52 weeks
Population: Our study was performed on an intention to treat basis. The number of participants in each included arm therefore was subsequently kept as the denominator at each follow - up regardless of any drop outs.
Measure: Number (99% Confidence Interval); unit: percentage of participants
Arm/Group | Control Group: Wait-and-see Treatment | Placebo Injection in Combination With Physical Therapy | Corticosteroid Injection in Combination With Physical Therapy
Number analyzed (Participants) | 60 | 58 | 59
percentage of participants
  6 weeks | 15 [3 to 27] | 24 [10 to 39] | 59 [43 to 76]
  12 weeks | 48 [32 to 65] | 45 [28 to 62] | 42 [26 to 59]
  26 weeks | 67 [51 to 82] | 69 [53 to 85] | 42 [26 to 59]
  52 weeks | 78 [65 to 92] | 78 [64 to 92] | 75 [60 to 89]

2. Secondary Outcome: Pain as Recorded by the Study Doctors on a Visual Analog Scale (VAS Scale)
Description: Pain in elbow as recorded by the study doctors on a 100 mm VAS-scale (Visual Analog Scale). The scale runs from 0 mm (no pain) to 100 mm (maximum pain), higher scores means worse outcome.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
mm | 29 (25) | 45 (23) | 44 (25)

3. Secondary Outcome: Pain as Recorded by the Study Doctors on a 100 mm VAS-scale (Visual Analog Scale).
Description: as for outcome 2
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
mm | 41 (26) | 33 (26) | 33 (26)

4. Secondary Outcome: Pain as Recorded by the Study Doctors on a 100 mm VAS-scale (Visual Analog Scale).
Description: as for outcome 2
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
mm | 38 (28) | 21 (22) | 19 (22)

5. Secondary Outcome: Pain as Recorded by the Study Doctors on a 100 mm VAS-scale
Description: as for outcome 2
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
mm | 19 (23) | 9 (11) | 13 (19)

6. Secondary Outcome: Pain-free Grip Strength Ratio
Description: Pain free grip strength registered with hand held dynamometer . Mean of three measurements as ratio of affected to unaffected side.Strength registered in kg. A ratio closer to zero signifies that pain occurs at the application of a small force signifying a more severe condition. A ratio approaching 1 signifies a milder complaint.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio x 100
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
Ratio x 100 | 58 (35) | 50 (29) | 57 (32)

7. Secondary Outcome: Pain-free Grip Strength Ratio
Description: Pain free grip strength registered with hand held dynamometer 30 31. Mean of three measurements as ratio of affected to unaffected side. Strength registered in kg. A ratio closer to zero signifies that pain occurs at the application of a small force signifying a more severe condition. A ratio approaching 1 signifies a milder complaint.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio x 100
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
Ratio x 100 | 64 (43) | 55 (25) | 63 (36)

8. Secondary Outcome: Pain-free Grip Strength Ratio
Description: Pain free grip strength registered with hand held dynamometer 30 31. Mean of three measurements as ratio of affected to unaffected side.Strength registered in kg. A ratio closer to zero signifies that pain occurs at the application of a small force signifying a more severe condition. A ratio approaching 1 signifies a milder complaint.
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio x 100
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
Ratio x 100 | 82 (48) | 76 (27) | 74 (37)

9. Secondary Outcome: Pain-free Grip Strength Ratio
Description: as for outcome 8
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio x 100
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
Ratio x 100 | 100 (33) | 90 (23) | 91 (23)

10. Secondary Outcome: Maximum Grip Strength Ratio
Description: Maximum grip strength registered with hand held dynamometer. Mean of three measurements as ratio of affected to unaffected side. Strength registered in kg. A ratio closer to zero signifies that pain hampers the application of grip force to a larger degree signifying a more severe condition. A ratio approaching 1 signifies a milder complaint where grip strength is not hampered by pain.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio x 100
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
Ratio x 100 | 87 (26) | 80 (25) | 74 (27)

11. Secondary Outcome: Maximum Grip Strength Ratio
Description: as for outcome 10
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio x 100
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
Ratio x 100 | 83 (29) | 88 (23) | 89 (28)

12. Secondary Outcome: Maximum Grip Strength Ratio
Description: as for outcome 10
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio x 100
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
Ratio x 100 | 89 (27) | 99 (20) | 99 (19)

13. Secondary Outcome: Maximum Grip Strength Ratio
Description: Maximum grip strength registered with hand held dynamometer. Mean of three measurements as ratio of affected to unaffected side.Strength registered in kg. A ratio closer to zero signifies that pain hampers the application of grip force to a larger degree signifying a more severe condition. A ratio approaching 1 signifies a milder complaint where grip strength is not hampered by pain.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio x 100
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
Ratio x 100 | 96 (19) | 102 (17) | 104 (15)

14. Secondary Outcome: Affected Function on 100 mm VAS-scale as Recorded by the Study Doctors
Description: To what extent is the use of the elbow affected registered on 100 mm VAS-scale. 0 mm represents use not affected. 100 mm signifies maximum affected function. Higher scores mean a worse outcome.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
mm | 25 (23) | 45 (24) | 38 (26)

15. Secondary Outcome: Affected Function on 100 mm VAS-scale as Recorded by the Study Doctors
Description: as for outcome 14
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
mm | 37 (29) | 32 (25) | 34 (28)

16. Secondary Outcome: Affected Function on 100 mm VAS-scale as Recorded by the Study Doctors
Description: as for outcome 14
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
mm | 28 (25) | 17 (22) | 16 (20)

17. Secondary Outcome: Affected Function on a 100 mm VAS-scale as Recorded by the Study Doctors
Description: as for outcome 14
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
mm | 16 (22) | 9 (15) | 10 (17)

18. Secondary Outcome: Overall Complaint on 100 mm VAS-scale as Recorded by the Study Doctors
Description: Overall complaint registered on VAS-scale as recorded by study doctors. 0 mm represents no overall complaint. 100 mm signifies maximum overall complaint. Higher scores mean a worse outcome.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
mm | 32 (26) | 50 (26) | 51 (28)

19. Secondary Outcome: Overall Complaint on 100 mm VAS-scale as Recorded by the Study Doctors
Description: as for outcome 18
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
mm | 43 (30) | 35 (28) | 36 (27)

20. Secondary Outcome: Overall Complaint on 100 mm VAS-scale as Recorded by the Study Doctors
Description: as for outcome 18
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
mm | 36 (26) | 19 (23) | 18 (20)

21. Secondary Outcome: Overall Complaint on 100 mm VAS-scale as Recorded by the Study Doctors
Description: as for outcome 18
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
mm | 20 (24) | 9 (13) | 12 (19)

22. Secondary Outcome: Pain Free Function Index of Everyday Activities
Description: Pain free function Index ( 0 - 8 ; 0: full function, 8 no function). Does the patient have pain on 8 every-day activities (dressing, eating, washing, household tasks, opening doors, carrying objects, with work, at sports). Recording a 0 on a complaint listed signifies full function, recording a 1 signifies no function. Thus the more activities with no function the higher score and the higher impairment.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
score on a scale | 2.78 (2.22) | 4.40 (2.01) | 4.82 (2.16)
Statistical Analysis 1: Comparison: Corticosteroid Injection in Combination With Physical Therapy vs Placebo Injection in Combination With Physical Therapy vs Control Group: Wait-and-see Treatment; Test type: Other; p < 0.01, linear generalized estimating equations; A linear GEE regression model adjusted for the significant covariates at p < 0.05 from the univariate GEE logistic regression models calculated for success
Statistical Analysis 2: Comparison: Corticosteroid Injection in Combination With Physical Therapy vs Placebo Injection in Combination With Physical Therapy vs Control Group: Wait-and-see Treatment; Test type: Other; p < 0.01, linear generalized estimating equations

23. Secondary Outcome: Pain Free Function Index of Everyday Activities
Description: as for outcome 22
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
score on a scale | 3.42 (2.63) | 3.62 (2.43) | 3.37 (2.36)

24. Secondary Outcome: Pain Free Function Index of Everyday Activities
Description: as for outcome 22
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
score on a scale | 2.97 (2.53) | 1.83 (2.08) | 2.00 (2.25)

25. Secondary Outcome: Pain Free Function Index of Everyday Activities
Description: as for outcome 22
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
score on a scale | 1.64 (2.04) | 1.03 (1.67) | 1.40 (1.90)

26. Secondary Outcome: No Pain on Three Point Likert Scale on Dorsiflexion of Wrist
Description: Percentage of patients reporting "no pain" on dorsiflexion of wrist on a three-point Likert scale on dorsiflexion of wrist. Scale: No pain - some pain - definite pain.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Number (99% Confidence Interval); unit: percentage of participants
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
percentage of participants | 36 [20 to 52] | 3 [-3 to 10] | 8 [-1 to 18]
Statistical Analysis 1: Comparison: Corticosteroid Injection in Combination With Physical Therapy vs Placebo Injection in Combination With Physical Therapy vs Control Group: Wait-and-see Treatment; Test type: Other; linear generalized estimating equations (GEE) regression model adjusted for significant covariates; between groups estimated odds ratio (OR) for no pain on two isometric movements using logistic GEE regression model adjusted for significant covariates; 99 % confidence intervals

27. Secondary Outcome: No Pain on Three Point Likert Scale on Dorsiflexion of Wrist
Description: as for outcome 26
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number (99% Confidence Interval); unit: percentage of patients
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
percentage of patients | 22 [8 to 36] | 12 [1 to 23] | 17 [4 to 29]

28. Secondary Outcome: No Pain on Three Point Likert Scale on Dorsiflexion of Wrist
Description: as for outcome 26
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Number (99% Confidence Interval); unit: percentage of patients
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
percentage of patients | 19 [6 to 32] | 29 [14 to 45] | 38 [22 to 54]

29. Secondary Outcome: No Pain on Three Point Likert Scale on Dorsiflexion of Wrist
Description: as for outcome 26
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Number (99% Confidence Interval); unit: percentage of patients
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
percentage of patients | 36 [20 to 52] | 60 [4 to 77] | 50 [33 to 67]

30. Secondary Outcome: No Pain on Three Point Likert Scale on Isometric Extension of Third Finger
Description: Percentage of patients reporting "no pain" on isometric extension of third finger on a three-point Likert scale on dorsiflexion of wrist. Scale: No pain - some pain - definite pain.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Number (99% Confidence Interval); unit: percentage of patients
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
percentage of patients | 44 [27 to 61] | 16 [3 to 28] | 17 [4 to 29]

31. Secondary Outcome: No Pain on Three Point Likert Scale on Isometric Extension of Third Finger
Description: as for outcome 30
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number (99% Confidence Interval); unit: percentage of patients
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
percentage of patients | 36 [20 to 52] | 24 [10 to 39] | 22 [8 to 35]

32. Secondary Outcome: No Pain on Three Point Likert Scale on Isometric Extension of Third Finger
Description: as for outcome 30
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Number (99% Confidence Interval); unit: percentage of patients
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
percentage of patients | 31 [15 to 46] | 53 [37 to 70] | 58 [42 to 75]

33. Secondary Outcome: No Pain on Three Point Likert Scale on Isometric Extension of Third Finger
Description: as for outcome 30
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Number (99% Confidence Interval); unit: percentage of patients
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Number analyzed (Participants) | 59 | 58 | 60
percentage of patients | 53 [36 to 69] | 76 [61 to 90] | 63 [47 to 79]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Corticosteroid Injection in Combination With Physical Therapy | Placebo Injection in Combination With Physical Therapy | Control Group: Wait-and-see Treatment
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/58 | 0/60
Other Adverse Events (participants affected / at risk) | 6/59 | 5/58 | 10/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Corticosteroid Injection in Combination With Physical Therapy (N=59) | Placebo Injection in Combination With Physical Therapy (N=58) | Control Group: Wait-and-see Treatment (N=60)
Increased pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
GI side effects (Gastrointestinal disorders) | 6 | 3 | 8
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Strict inclusion criteria limit generalizability.The patients were not blinded to physiotherapy.Home exercises not logged.Only one physiotherapist.No individual adjustment of treatment. .We did not look specifically at recurrence rates.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes